CLINICAL TRIAL: NCT06087458
Title: Phase 1/2a Dose Escalation Study of VOY-101 in Patients With Advanced Non- Neovascular Age-Related Macular Degeneration
Brief Title: Study of VOY-101 in Patients With Advanced Non-Neovascular Age-Related Macular Degeneration
Acronym: JOURNEY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perceive Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI-AMD-002
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy; Non-neovascular AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Phase 1 follows a standard dose escalation model to evaluate safety and tolerability of VOY-101 and recommended Phase 2a dose (RP2D). This dose will be used in Phase 2a to evaluate the safety and efficacy of VOY-101 in the study eye compared to untreated fellow eye.
Masking Description: Central Reading Center is masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VOY-101 (Experimental): Single intravitreal injection of VOY-101
  Interventions: Biological: VOY-101
- Controll (No Intervention): Fellow Eye

INTERVENTIONS:
Biological: VOY-101 — VOY-101
  Arms: VOY-101

SUMMARY:
The Phase 1 safety study of VOY-101 comprises of escalating dose Cohorts, followed by a Phase 2a.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center Phase 1/2a study to evaluate the safety of a single, unilateral intravitreal (IVT) injection of escalating dose levels of VOY-101 therapy in subjects with advanced non-neovascular age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Are ≥60 years of age at the time of consent.
* Are willing and able to understand and provide written informed consent.
* Are willing and able to return for scheduled treatment and follow-up examinations.
* Are able to undergo ETDRS BCDVA testing and ophthalmic imaging.
* Well-demarcated GA secondary to AMD in the absence of MNV and in the absence of history of MNV for both eyes.
* Absence of signs of non-exudative MNV.
* Additional Ocular Inclusion Criteria for both eyes.
* Meet certain genotype criteria for risk of AMD.

Exclusion Criteria:

* Are women of childbearing potential (WOCBP) and are pregnant or unwilling to use and document use of effective contraception for the duration of the study.
* Additional Systemic, Ocular, and Genetic Exclusion Criteria.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall effect of treatment on retinal structural health | Week 48
  GA growth rate and Change in Ellipsoid Zone Integrity

SECONDARY OUTCOMES:
Overall effect of treatment on retinal structural health | Weeks 36, 48, and 96
  GA Growth Rate and Change in Ellipsoid Zone Integrity
Effect of treatment on vision function | Change from baseline
  Change from Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) BCDVA and LLVA and microperimetry.
Incidence of neovascular AMD | Baseline to Week 96
  Incidence, frequency, severity, and timing of development of neovascular AMD
VOY-101 Safety | Baseline to Week 96
  Frequency of related ocular and systemic AEs (SAEs and non-serious), adverse events of special interest (AESI) and non-serious TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fung, MD, Study Director — Perceive Biotherapeutics, Inc.
Locations (11):
- United States (7):
  - Retina Macula Institute of AZ, Scottsdale, Arizona
  - The Retina Partners, Encino, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Retina Consultants San Diego, San Diego, California
  - Star Retina, Burleson, Texas
  - Retina Center of Texas, Southlake, Texas
  - University of Utah John A. Moran Eye Center, Salt Lake City, Utah
- Australia (2):
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Cerulea Clinical Trials, East Melbourne, Victoria
- Israel (2):
  - Rambam Medical Center, Haifa
  - Tel-Aviv Sourasky Medical Center, Ophthalmology Division, Tel Aviv

IPD SHARING:
Plan to Share IPD: No